CLINICAL TRIAL: NCT06422221
Title: An Oral Doxycycline Regimen to Prevent Bacteremia Following Dental Procedures
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Collaborators: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Pedro DIz DIos, Full Professor, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Doxycycline Regimen
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Bacteremia; Endocarditis
MeSH Terms: conditions — Bacteremia; Endocarditis | interventions — Clindamycin; Doxycycline

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Intervention (No Intervention): Receiving no prophylaxis
- Clindamycin (Active Comparator): Receiving 600 mg oral Clindamycin 1 hour before general anesthesia and before any dental manipulation
  Interventions: Drug: Clindamycin
- Doxycycline (Active Comparator): Receiving 100 mg oral Doxycycline 1 hour before general anesthesia and before any dental manipulation
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Clindamycin — Receiving 600 mg oral Clindamycin 1 hour before general anesthesia and before any dental manipulation
  Arms: Clindamycin
Drug: Doxycycline — Receiving 100 mg oral Doxycycline 1 hour before general anesthesia and before any dental manipulation
  Arms: Doxycycline

SUMMARY:
Although controversy exists regarding the efficacy of antibiotic prophylaxis for patients at risk of infective endocarditis, expert committees continue to publish recommendations for antibiotic prophylactic regimens. The last American Heart Association (AHA) and European Society of Cardiology (ESC) guidelines include several important changes, highlighting that clindamycin (CLI) is no longer recommended as an alternative to amoxicillin in those allergic to penicillin. This new project aims to evaluate the effectiveness of oral doxycycline in preventing post-dental extraction bloodstream infection.

DETAILED DESCRIPTION:
PURPOSE: Despite the controversy about the risk of developing bacterial endocarditis of oral origin, numerous Expert Committees in different countries continue to publish prophylactic regimens. To date, the literature is unclear about the role of antimicrobial prophylaxis in the prevention of bacteremia following dental procedures. The aim of this study is to evaluate the efficacy of prophylactic dosage with oral doxycycline (DXC) in the prevention of bacteremia following dental extractions.

SELECTION OF THE STUDY GROUP AND STUDY DESIGN: The study group will comprise patients who, for behavioral reasons (autism, learning disabilities, phobias, etc.), will undergo dental extractions under general anesthesia in the Santiago de Compostela University Hospital (Santiago de Compostela, Spain). 150 patients will be selected and will be randomly distributed into 3 study groups: control group (receiving no prophylaxis), CLI group (receiving 600 mg oral CLI) and DXC group (receiving 100 mg oral DXC).

COLLECTION OF SAMPLES FOR BLOOD CULTURE: To determine the prevalence of bacteremia, a peripheral venous blood sample (10 ml) will be drawn from each patient. Samples will be inoculated in BACTEC plus (Becton Dickinson and Company, Sparks, MD) aerobic and anaerobic blood culture bottles, and will be processed in the Bactec 9240 (Becton Dickinson).

MICROBIOLOGICAL ANALYSIS OF BLOOD CULTURES: A Gram stain will be performed on each positive blood culture. The positive blood cultures in the aerobic media will be subcultured on blood agar and chocolate agar in an atmosphere of 5 to 10% carbon monoxide and on MacConkey agar under aerobic conditions. The same protocol will be used for the positive blood cultures in the anaerobic media, with subculture on Schaedler agar and incubation in an anaerobic atmosphere. The bacteria isolated will be identified by using the battery of biochemical tests provided with the Vitek system for Gram-positive bacteria, Neisseria spp., Haemophilus spp., and obligate anaerobic bacteria. The viridans group streptococci will be classified into five groups, the Streptococcus mitis, S. anginosus, S. salivarius, S. mutans, and S. bovis groups, by applying the Ruoff criteria. Facklam's criteria will be used to identify unusual Streptococcus spp. and other Gram-positive cocci in chains.

The subculture and further identification of the isolated bacteria will be performed by conventional microbiological techniques. The collection, handling, and transport of the blood samples for blood culture will be performed according to the recommendations of the Spanish Society of Infectious Diseases and Clinical Microbiology.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have at least 10 teeth.
* Subjects must have the need for a dental extraction under general anesthesia (for behavioral reasons).
* Subjects will be recruited regardless of the extent and severity of their dental and/or periodontal disease.

Exclusion Criteria:

* Age under 18 years
* Body weight under 40 kg
* Receipt of antibiotics in the previous 3 months
* Routine use of oral antiseptics
* A history of allergy or intolerance to doxycycline
* A history of allergy or intolerance to cindamycin
* Any type of congenital or acquired immunodeficiency
* Any known risk factor for bacterial endocarditis
* Any known risk factor for prolonged bleeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Bacteremia in participants receiving a prophylactic dosage with oral doxycyclin | Changes from baseline at 30 seconds and 15 minutes after the final dental extraction
  Positive cultures

SECONDARY OUTCOMES:
Bacteremia in participants receiving a prophylactic dosage with oral clindamycin | Changes from baseline at 30 seconds and 15 minutes after the final dental extraction
  Positive cultures
Bacteremia in participants receiving no prophylaxis | Changes from baseline at 30 seconds and 15 minutes after the final dental extraction
  Positive cultures

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Diz Dios, Principal Investigator — Santiago de Compostela University
Locations (1):
- Santiago de Compostela University Hospital, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available on request
Supporting Information: CSR
Time Frame: By the end of the study (for 1 year)
Access Criteria: On request

REFERENCES:
- [Background] Diz Dios P. Infective endocarditis prophylaxis. Oral Dis. 2014 May;20(4):325-8. doi: 10.1111/odi.12221. Epub 2014 Jan 13. PMID 24373017
- [Background] Valdes C, Tomas I, Alvarez M, Limeres J, Medina J, Diz P. The incidence of bacteraemia associated with tracheal intubation. Anaesthesia. 2008 Jun;63(6):588-92. doi: 10.1111/j.1365-2044.2008.05449.x. PMID 18477269
- [Background] Pineiro A, Tomas I, Blanco J, Alvarez M, Seoane J, Diz P. Bacteraemia following dental implants' placement. Clin Oral Implants Res. 2010 Sep;21(9):913-8. doi: 10.1111/j.1600-0501.2010.01928.x. PMID 20701619
- [Background] Diz Dios P, Tomas Carmona I, Limeres Posse J, Medina Henriquez J, Fernandez Feijoo J, Alvarez Fernandez M. Comparative efficacies of amoxicillin, clindamycin, and moxifloxacin in prevention of bacteremia following dental extractions. Antimicrob Agents Chemother. 2006 Sep;50(9):2996-3002. doi: 10.1128/AAC.01550-05. PMID 16940094
- [Background] Limeres Posse J, Alvarez Fernandez M, Fernandez Feijoo J, Medina Henriquez J, Lockhart PB, Chu VH, Diz Dios P. Intravenous amoxicillin/clavulanate for the prevention of bacteraemia following dental procedures: a randomized clinical trial. J Antimicrob Chemother. 2016 Jul;71(7):2022-30. doi: 10.1093/jac/dkw081. Epub 2016 Mar 29. PMID 27029851
- [Background] Relvas M, Diz P, Seoane J, Tomas I. Oral Health Scales: design of an oral health scale of infectious potential. Med Oral Patol Oral Cir Bucal. 2013 Jul 1;18(4):e664-70. doi: 10.4317/medoral.18427. PMID 23524418
- [Background] Martins CC, Lockhart PB, Firmino RT, Kilmartin C, Cahill TJ, Dayer M, Occhi-Alexandre IGP, Lai H, Ge L, Thornhill MH. Bacteremia following different oral procedures: Systematic review and meta-analysis. Oral Dis. 2024 Apr;30(3):846-854. doi: 10.1111/odi.14531. Epub 2023 Mar 29. PMID 36750413
- [Background] Thornhill MH, Gibson TB, Yoon F, Dayer MJ, Prendergast BD, Lockhart PB, O'Gara PT, Baddour LM. Endocarditis, invasive dental procedures, and antibiotic prophylaxis efficacy in US Medicaid patients. Oral Dis. 2024 Apr;30(3):1591-1605. doi: 10.1111/odi.14585. Epub 2023 Apr 27. PMID 37103475
- [Background] Diniz Freitas M, Alvarez Fernandez M, Vasallo Vidal FJ, Limeres Posse J, Diz Dios P, Fernandez Feijoo J. Oral amoxicillin/clavulanate for the prevention of bacteremia following dental extractions. Oral Dis. 2023 Jul;29(5):2272-2276. doi: 10.1111/odi.14221. Epub 2022 May 13. PMID 35467064
- [Background] Dayer MJ, Jones S, Prendergast B, Baddour LM, Lockhart PB, Thornhill MH. Incidence of infective endocarditis in England, 2000-13: a secular trend, interrupted time-series analysis. Lancet. 2015 Mar 28;385(9974):1219-28. doi: 10.1016/S0140-6736(14)62007-9. Epub 2014 Nov 18. PMID 25467569
- [Background] Lean SSH, Jou E, Ho JSY, Jou EGL. Prophylactic antibiotic use for infective endocarditis: a systematic review and meta-analysis. BMJ Open. 2023 Aug 22;13(8):e077026. doi: 10.1136/bmjopen-2023-077026. PMID 37607797
- [Background] Dayer MJ, Thornhill M, Baddour LM. Antibiotic prophylaxis for patients at risk of infective endocarditis: an increasing evidence base? Br J Cardiol. 2023 Feb 21;30(1):6. doi: 10.5837/bjc.2023.006. eCollection 2023. PMID 37705833